CLINICAL TRIAL: NCT03276143
Title: A Randomized, Active-comparator-controlled, Multicenter Study to Assess the Safety and Efficacy of Different Doses of BAY1213790 for the Prevention of Venous Thromboembolism in Patients Undergoing Elective Primary Total Knee Arthroplasty, Open-label to Treatment and Observer-blinded to BAY1213790 Doses
Brief Title: FactOr XIa inhibiTion for the pRevention of venOus Thromboembolism in Patients Undergoing Total Knee Arthroplasty
Acronym: FOXTROT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17664; 2016-002681-31 (EudraCT Number)
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Knee Arthroplasty, Total
Keywords: Orthopedic surgery; Venous thromboembolism; Deep vein thrombosis (DVT); Anticoagulation
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis | interventions — Enoxaparin; apixaban; osocimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Enoxaparin (Active Comparator): Adult patients who underwent Total Knee Arthroplasty (TKA) surgery and received enoxaparin for at least 10 days until venography was performed.
  Interventions: Drug: Enoxaparin
- Apixaban (Active Comparator): Adult patients who underwent Total Knee Arthroplasty (TKA) surgery and received apixaban for at least 10 days until venography was performed.
  Interventions: Drug: Apixaban
- BAY1213790 0.3 mg/kg (post-surgery) (Experimental): Adult patients who underwent Total Knee Arthroplasty (TKA) surgery and received 0.3 mg BAY1213790 once post-surgery.
  Interventions: Drug: BAY1213790
- BAY1213790 0.6 mg/kg (post-surgery) (Experimental): Adult patients who underwent Total Knee Arthroplasty (TKA) surgery and received 0.6 mg BAY1213790 once post-surgery.
  Interventions: Drug: BAY1213790
- BAY1213790 1.2 mg/kg (post-surgery) (Experimental): Adult patients who underwent Total Knee Arthroplasty (TKA) surgery and received 1.2 mg BAY1213790 once post-surgery.
  Interventions: Drug: BAY1213790
- BAY1213790 1.8 mg/kg (post-surgery) (Experimental): Adult patients who underwent Total Knee Arthroplasty (TKA) surgery and received 1.8 mg BAY1213790 once post-surgery.
  Interventions: Drug: BAY1213790
- BAY1213790 0.3 mg/kg (pre-surgery) (Experimental): Adult patients who underwent Total Knee Arthroplasty (TKA) surgery and received 0.3 mg BAY1213790 once pre-surgery.
  Interventions: Drug: BAY1213790
- BAY1213790 1.8 mg/kg (pre-surgery) (Experimental): Adult patients who underwent Total Knee Arthroplasty (TKA) surgery and received 1.8 mg BAY1213790 once pre-surgery.
  Interventions: Drug: BAY1213790

INTERVENTIONS:
Drug: Enoxaparin — 40 mg enoxaparin administered as subcutaneous injection once daily
  Arms: Enoxaparin
Drug: Apixaban — 2.5 mg apixaban administered as tablet orally twice daily
  Arms: Apixaban
Drug: BAY1213790 — Single dose of BAY1213790 administered as intravenous infusion
  Other Names: Osocimab
  Arms: BAY1213790 0.3 mg/kg (post-surgery); BAY1213790 0.3 mg/kg (pre-surgery); BAY1213790 0.6 mg/kg (post-surgery); BAY1213790 1.2 mg/kg (post-surgery); BAY1213790 1.8 mg/kg (post-surgery); BAY1213790 1.8 mg/kg (pre-surgery)

SUMMARY:
This study was to compare the study drug BAY1213790 to existing therapies, i.e. enoxaparin or apixaban, for the prevention of blood clotting and safety in patients undergoing total knee arthroplasty (TKA). The study was open-label, but observer-blinded for the different doses of BAY1213790. This means that it was known which treatment was given, but it was not known which dose of BAY1213790 was administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years and undergoing elective primary, unilateral Total Knee Arthroplasty (TKA)
* Women of non-childbearing potential

Exclusion Criteria:

* High risk for clinically significant bleeding
* Prior deep vein thrombosis
* Body weight above 135 kg
* Creatinine clearance below 60 ml/min
* Recent (<6 months) myocardial infarction or ischemic stroke
* Contraindication listed in the local label of the comparator treatments
* Requirement for full dose anticoagulation or dual antiplatelet therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 813 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
Incidence of composite endpoint consisting of asymptomatic DVT as detected by mandatory bilateral venography, objectively confirmed symptomatic DVT, non-fatal PE, fatal PE, unexplained death for which PE cannot be excluded | Up to 15 days
  DVT - Deep vein thrombosis / PE - Pulmonary embolism All suspected events were reviewed and classified by the Central Independent Adjudication Committee.
Incidence of composite endpoint of major and clinically relevant non-major bleeding | Up to 15 days
  All suspected events were reviewed and classified by the Central Independent Adjudication Committee.

SECONDARY OUTCOMES:
Incidence of composite endpoint of symptomatic DVT, non-fatal PE, fatal PE, unexplained death for which PE cannot be excluded up to Day 157 or objectively confirmed asymptomatic DVT up to Day 15 | Up to 157 days
  All suspected events were reviewed and classified by the Central Independent Adjudication Committee.
Incidence of composite endpoint of major and clinically relevant non-major bleeding | Up to 157 days
  All suspected events were reviewed and classified by the Central Independent Adjudication Committee.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (54):
- Bulgaria (3):
  - UMHAT Sveti Georgi, Plovdiv
  - Acibadem City Clinic Multiprofile Hospital for Active Treatm, Sofia
  - UMHAT Tsaritsa Joanna-ISUL EAD Sofia, Sofia
- Medical Investigative & Clinical Evaluation Inc., Windsor, Ontario, Canada
- Czechia (4):
  - Fakultni nemocnice u sv. Anny, Brno
  - Nemocnice Ceske Budejovice, a.s., České Budějovice
  - Okresni nemocnice Jindrichuv Hradec, Jindřichův Hradec
  - Regional Hospital Pardubice, Pardubice
- Greece (4):
  - KAT General Hospital of Athens, Kifissia
  - Konstantopoulio General Hospital of Nea Ionia - Agia Olga, Nea Ionia
  - University General Hospital of Patras, Pátrai
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- Israel (5):
  - Rambam Health Corporation, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Clalit Health Services through Rabin Medical Center - Beilinson Campus, Petah Tikva
  - Kaplan Medical Center, Rehovot
- Latvia (4):
  - Liepaja Regional Hospital, Liepāja
  - Riga 2nd City Hospital, Riga
  - Hospital of Traumatology and Orthopaedics, Riga
  - Valmiera Hospital, Valmiera
- Lithuania (5):
  - Kaunas clinical hospital (Laisves ave.), Kaunas
  - Lithuanian university of Health science, Kaunas
  - PI Klaipedos University Hospital, Klaipėda
  - Republican Vilnius University Hospital, Vilnius
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Poland (6):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Wojewódzki Szpital Zespolony, Kielce
  - Szpital Specjalistyczny im. Rydygiera, Krakow
  - Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi, Lodz
  - Wojewodzki Szpital Specjalistyczny im. S. Wyszynskiego SPZOZ, Lublin
  - Uniwersytecki Szpital Kliniczny UM we Wroclawiu, Wroclaw
- Portugal (5):
  - Hospital de Cascais, Alcabideche, Lisbon District
  - CHS - Hospital Ortopedico Sant Iago do Outao, Setúbal, Setúbal District
  - CHBV - Hospital Infante D. Pedro, Aveiro
  - CHL - Hospital Santo Andre, Leiria
  - ULSAM - Hospital Santa Luzia, Viana do Castelo
- Russia (5):
  - Russian Scientific Center n.a. acad. G.A. Ilizarov, Kurgan
  - Privolzhskiy Federal Medical Research Center, Nizhny Novgorod
  - City Hospital #2, Saint Petersburg
  - Sci-Res. Institute of Traumatology and Orthopaedia, Saint Petersburg
  - Clinical Hospital for Emergency Care n.a. N.V.Solovyov, Yaroslavl
- South Africa (3):
  - Pretoria Academic Hospital New, Pretoria, Gauteng
  - UCT Clinical Research Centre, Cape Town, Western Cape
  - Clinical Projects Research SA, Worcester, Western Cape
- Spain (6):
  - Ciutat Sanitària i Universitària de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Fundación Hospital Alcorcón, Alcorcón, Madrid
  - Ciutat Sanitària i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Clínico Universitario San Carlos, Madrid
- Ukraine (3):
  - Cherkasy Reg Clinical Hospital of Cherkasy Reg Council, Cherkasy
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - Kyiv Regional Clinical Hospital, Kyiv

REFERENCES:
- [Derived] Weitz JI, Bauersachs R, Becker B, Berkowitz SD, Freitas MCS, Lassen MR, Metzig C, Raskob GE. Effect of Osocimab in Preventing Venous Thromboembolism Among Patients Undergoing Knee Arthroplasty: The FOXTROT Randomized Clinical Trial. JAMA. 2020 Jan 14;323(2):130-139. doi: 10.1001/jama.2019.20687. PMID 31935028